CLINICAL TRIAL: NCT03695432
Title: Role of Probiotic and Influenza Vaccination on Immune Response Enchancement and Influenza-Like Illness Incidence Reduction in Elderly
Brief Title: Probiotic and Influenza Vaccination to Reducing Influenza-like Illness Incident in Elderly
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Sukamto Koesnoe, Principal investigator, Indonesia University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: Vaccine2016
Record Dates: First submitted 2018-09-28; First posted 2018-10-04 (Actual); Last update posted 2018-10-05 (Actual); Status verified 2018-10

CONDITIONS: Influenza-like Illness
Keywords: Influenza; Vaccine; Probiotic; Influenza-like Illness
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (4):
- Vaccine (Experimental): Flubio (A/California/7/2009, A/Texas/50/2012 and B/Massachusetts/2/2012) Vaccine 0,5 ml for every subjects The vaccine will be given intramuscularly
  Interventions: Biological: Flubio
- Probiotic (Experimental): Lacidofil (Lactobacillus acidophilus Rossel-52 and Lactobacillus rhamnosus Rosell-11 with maltodextrin 211 mg, magnesium stearat 8 mg and ascorbic acid 1 mg) antibiotic
  Interventions: Dietary Supplement: Lacidofil
- Placebo Vaccine (Placebo Comparator): Nacl 0,9% 0,5 ml The placebo vaccine will be given intramuscularly
  Interventions: Other: Placebo Vaccine
- Placebo probiotic (Placebo Comparator): capsul
  Interventions: Other: Placebo probiotic

INTERVENTIONS:
Biological: Flubio — Flubio (A/California/7/2009, A/Texas/50/2012 and B/Massachusetts/2/2012) Vaccine 0,5 ml for every subjects The vaccine will be given intramuscularly
  Arms: Vaccine
Dietary Supplement: Lacidofil — Lacidofil (Lactobacillus acidophilus Rossel-52 and Lactobacillus rhamnosus Rosell-11 with maltodextrin 211 mg, magnesium stearat 8 mg and ascorbic acid 1 mg) antibiotic The antibiotic will be given 2 times each day for 6 months
  Arms: Probiotic
Other: Placebo Vaccine — Nacl 0,9% 0,5 ml The placebo vaccine will be given intramuscularly
  Arms: Placebo Vaccine
Other: Placebo probiotic — Capsul
  Arms: Placebo probiotic

SUMMARY:
To asses the effect of the probiotic and influenza vaccination alone and combination on enhancing immune response to influenza-like illness (ILI) and reducing ILI incidence in the elderly

DETAILED DESCRIPTION:
To see percetange of subjects seroconvertion and seroprotection before and after intervention in the elderly (>60 years), and monitored for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* all health elderly aged ≥ 60 years
* who came to the vaccination and health education activities in the entire East Jakarta District Health Center
* with Body Mass Index (BMI) 17,5-29,9
* healthy mental status (MMSE score of 28-30)

Exclusion Criteria:

* subject who have contraindications to influenza vaccinations
* are undergoing treatment related to immune system modulation in the past 4 weeks
* therapy for immunossuppresants and/ or corticosteroids eqivalent to prednisone ≥ 20 mg/day that is being lived more than 2 weeks or has only been stopped less than 3 months before the study
* recieved influenza vaccination less than one year before
* Currently consuming probiotic agents, either in the form of a manufacturer or natural for more than 7 days.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 910 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2015-04 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
The precentage enhancement of the immune response to flubio vaccine and probiotic compared to plasebo 6 months after vaccination | 6 months

SECONDARY OUTCOMES:
Percentage of subjects with anti HI titer >=1:40 | 6 months
  Describe seroprotection on 4-weeks, 4-months, and 6-months after interventions in elderly
Percentage subjects with increasing antibody titer >=4 times | 6 months
  Describe seroconvertion on 4-weeks, 4-months, and 6-months after interventions in elderly

CONTACTS AND LOCATIONS:
Overall Officials: Sukamto Koesnoe, MD, Principal Investigator — Division of Allergic and Imunologic, Department of Internal Medicine, Indonesia University
Locations (1):
- Integrated Health Post, at Pulo Gadung District, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Koesnoe S, Masjkuri N, Adisasmita A, Djauzi S, Kartasasmita C, Sundoro J, Nadjib M, Korib M, Muthia AN, Muzellina VN, Habibah U, Nursyirwan SA, Djaya KH, Bachtiar NS, Sari RM. A randomized controlled trial to evaluate the effect of influenza vaccination and probiotic supplementation on immune response and incidence of influenza-like illness in an elderly population in Indonesia. PLoS One. 2021 Dec 16;16(12):e0250234. doi: 10.1371/journal.pone.0250234. eCollection 2021. PMID 34914726